CLINICAL TRIAL: NCT05591222
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Trial to Investigate the Efficacy and Safety of Daxdilimab Subcutaneous Injection in Reducing Disease Activity in Adult Participants With Moderate-to-Severe Primary Discoid Lupus Erythematosus
Brief Title: Study of Daxdilimab (HZN-7734) in Participants With Moderate-to-Severe Primary Discoid Lupus Erythematosus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor business decision, not related to safety concerns.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HZNP-DAX-202; 2023-509746-35-00 (EU CTIS Number)
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Discoid Lupus Erythematosus
Keywords: Discoid Lupus Erythematosus; Immune System Diseases; Lupus Erythematosus, Cutaneous; Skin Diseases; Connective Tissue Diseases
MeSH Terms: conditions — Lupus Erythematosus, Discoid; Immune System Diseases; Lupus Erythematosus, Cutaneous; Skin Diseases; Connective Tissue Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Administration of placebo Q4W from Day 1 through Week 20.
  Interventions: Drug: Placebo
- Daxdilimab; Low Dose (Experimental): Administration of daxdilimab low dose Q4W from Day 1 through Week 20.
  Interventions: Drug: Daxdilimab
- Daxdilimab; High Dose (Experimental): Administration of daxdilimab high dose Q4W from Day 1 through Week 20.
  Interventions: Drug: Daxdilimab

INTERVENTIONS:
Drug: Placebo — Placebo will be administered subcutaneously as two injections for each dose.
  Arms: Placebo
Drug: Daxdilimab — Daxdilimab will be administered subcutaneously as two injections for each dose.
  Other Names: HZN-7734
  Arms: Daxdilimab; High Dose; Daxdilimab; Low Dose

SUMMARY:
A Phase 2, double-blind, randomized, placebo-controlled parallel-group study to evaluate the efficacy and safety of daxdilimab in participants with moderate-to-severe active primary Discoid Lupus Erythematosus (DLE) refractory to standard of care.

DETAILED DESCRIPTION:
Approximately 72 participants will be enrolled to receive daxdilimab or placebo administered subcutaneously once every four weeks (Q4W) from Day 1 to Week 20. The maximum trial duration per participant is approximately 36 weeks including screening, the 24 weeks for the treatment period where participants will receive daxdilimab or placebo, and approximately 8 weeks for the follow-up period. Safety evaluations will be performed regularly throughout the course of the study.

Acquired from Horizon in 2024.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to understand and provide written informed consent.
* Willing and able to comply with the prescribed treatment protocol and evaluations for the duration of the trial.
* A diagnosis of DLE for ≥ 6 months prior to screening supported by a history of:

  1. A biopsy or
  2. a clinical feature score of ≥ 7 on the DLE Classification Criteria (DLECC) scale.
* Currently active discoid lupus with all the following:

  1. Digital photography adjudicated with central reading to confirm a currently active discoid disease lesion.
  2. CLASI-A score ≥ 8 related to discoid lesions at Baseline.
* Treatment refractory DLE defined as active disease despite current or historical treatment with a systemic treatment.
* Females are eligible to participate if they are not pregnant or breastfeeding, and meet the contraceptive/barrier requirement(s).
* Males are eligible to participate if they agree to the contraceptive/barrier requirement(s).
* Vaccination status should be up to date per local standards.

Key Exclusion Criteria:

* Participation in another clinical study with an investigational drug within 4 weeks prior to Randomization or within 5 published half-lives, whichever is longer.
* Any condition that, in the opinion of the Investigator, would interfere with evaluation of the investigational product (IP) or interpretation of participant safety or trial results.
* Weight > 160 kg (352 pounds) at Screening.
* History of allergy, hypersensitivity reaction, or anaphylaxis to any component of the IP or to a previous monoclonal antibody (mAb) or human immunoglobin (Ig) therapy.
* Breastfeeding or pregnant women or women who intend to become pregnant anytime from signing the informed consent form (ICF) through 6 months after receiving the last dose of IP.
* Splenectomy.
* Spontaneous or induced abortion, still or live birth, or pregnancy ≤ 4 weeks prior to screening through randomization.
* History of clinically significant cardiac disease including unstable angina, myocardial infarction, congestive heart failure within 6 months prior to Randomization; arrhythmia requiring active therapy, except for clinically insignificant extra systoles, or minor conduction abnormalities.
* History of cancer within the past 5 years, except as follows:

  * Cutaneous basal cell or squamous cell carcinoma treated with curative therapy.
* Any underlying condition that in the opinion of the Investigator significantly predisposes the participant to infection.
* Known history of a primary immunodeficiency or an underlying condition, such as known human immunodeficiency virus (HIV) infection, or a positive result for HIV infection per central laboratory.
* Participants with positive hepatitis B serologic test results.
* All participants will undergo testing for hepatitis C antibody (HCVAb) during Screening.
* Participants who are HCVAb positive will be reflex tested for hepatitis C virus (HCV) RNA and if HCV RNA is positive, the participant is not eligible for the study.
* Active tuberculosis (TB), or a positive interferon-gamma release assay (IGRA) test at screening, unless documented history of appropriate treatment for active or latent TB.

Participants with an indeterminate IGRA test result can repeat the test, but if the repeat test is also indeterminate, they will be excluded.

* Any severe herpes virus family infection (including Epstein-Barr virus, cytomegalovirus (CMV)) at any time prior to Randomization, including, but not limited to, disseminated herpes, herpes encephalitis, recent recurrent herpes zoster (defined as 2 episodes within the last 2 years), or ophthalmic herpes.
* Any herpes zoster, CMV, or Epstein-Barr virus infection that was not completely resolved 12 weeks prior to Randomization.
* Opportunistic infection requiring hospitalization or parenteral antimicrobial treatment within 2 years prior to Randomization.
* Any acute illness or evidence of clinically significant active infection on Day 1.
* Participants who have COVID-19 or other significant infection, or in the judgment of the Investigator, may be at a high risk of COVID-19 or its complications should not be randomized.
* Systemic lupus erythematosus defined by fulfilling 2020 American College of Rheumatology/European Alliance of Associations for Rheumatology criteria for systemic lupus erythematosus (SLE).
* Current diagnosis of a systemic connective tissue disease.
* Current inflammatory skin disease other than DLE, that, in the opinion of the Investigator, could interfere with the inflammatory skin assessments and confound the disease activity assessments.
* Exposure to an experimental drug either 30 days, 5 half-lives of the agent, or twice the duration of the biological effect of the agent, whichever is longer, prior to Randomization and through the final trial visit.
* Receipt of a live-attenuated vaccine within 4 weeks prior to Randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Mean Change in Cutaneous Lupus Erythematosus Disease and Severity Index-Activity (CLASI-A) Score from Baseline to Week 24 | Baseline to Week 24

SECONDARY OUTCOMES:
Percentage of Participants who Achieve 0 or 1 on the Cutaneous Lupus Activity-investigator's Global Assessment (CLA-IGA) scale at Week 24 | Week 24
  CLA-IGA will be assessed by 5-point Likert Scale (0-4).
Percentage of Participants who Achieve a ≥ 50% Reduction in CLASI-A Score from Baseline at Week 24 | Baseline to Week 24
Mean Change in the Score of Activity and Damage in Discoid Lupus Erythematosus (SADDLE) from Baseline to Week 24 | Baseline to Week 24
Serum Concentration of Daxdilimab Over Time | Day 1 to Week 24
Percentage of Participants who Develop Anti-Drug Antibodies (ADA) | Day 1 to Week 32
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Day 1 to SFU2 (Week 32)
  AEs, Serious AEs (SAEs) and AEs of Special Interest (AESIs) will be monitored. An AE is any untoward medical occurrence in a clinical trial participant, temporally associated with the use of trial intervention, whether or not considered related to the trial intervention.
  An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria listed:
  1. Results in death
  2. Is life-threatening. An AESI is an AE of scientific and medical interest specific to understanding of the IP and may require close monitoring and collection of additional information by the Investigator. An AESI may be serious or nonserious.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (68):
- United States (16):
  - Arkansas Research Trials, North Little Rock, Arkansas
  - Wallace Medical Group, Beverly Hills, California
  - The Center for Dermatology Clinical Research, Fremont, California
  - Clinical Science Institute, Santa Monica, California
  - Miami Dermatology & Laser Research, Miami, Florida
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Detroit Clinical Research Center, PC, Farmington Hills, Michigan
  - Michigan Dermatology Institute, Waterford, Michigan
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Forest Hills Dermatology, Forest Hills, New York
  - Ohio State University, Columbus, Ohio
  - Wright State Physicians, Fairborn, Ohio
  - Paddington Testing Company, Inc., Philadelphia, Pennsylvania
  - Autoimmune Skin Diseases Unit, Dept. of Dermatology, Philadelphia, Pennsylvania
  - Center for Clinical Studies (Cypress), Houston, Texas
- Argentina (2):
  - Fundacion Scherbovsky, Mendoza, Mendoza Province
  - CIPREC, Ciudad Autonoma Buenos Aires
- Brazil (14):
  - HUWC - UFC - Hospital Universitário Walter Cantídio - Universidade Federal do Ceará, Fortaleza, Ceará
  - Hospital Universitário Evangélico Mackenzie, Água Verde, Paraná
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, CIP - Centro Integrado de Pesquisa, Sao Jose Rio, Preto Sao Paulo
  - Complexo Hospitalar de Niterói, Niterói, Rio Do Janeiro
  - Instituto Brasil de Pesquisa Clínica-IBPCLIN S/A, Rio de Janeiro, Rio Do Janeiro
  - Fundação Universidade de Caxias do Sul - Instituto de Pesquisas em Saúde da Universidade de Caxias do Sul, Caxias do Sul, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - LMK Serviços Médicos S/S, Porto Alegre, Rio Grande do Sul
  - Universidade Estadual de Campinas, Campinas, São Paulo
  - Hospital Christovão da Gama - Centro de Estudos, Santo André, São Paulo
  - Centro Multidisciplinar de Estudos Clinicos, São Bernardo do Campo, São Paulo
  - IMC - Instituto de Moléstias Cardiovasculares Tatuí, Tatuí, São Paulo
  - IPITEC Instituto de Pesquisa Inovação Tecnológica, São Paulo
- Bulgaria (4):
  - DCC 'Sveti Georgi' EOOD, Haskovo
  - Ambulatory for specialized medical care - individual practice for specialized medical care - skin and venereal diseases, Sofia
  - DCC "Alexandrovska" EOOD, Sofia
  - Medical Center Eurohealth EOOD, Sofia
- Canada (5):
  - Alberta DermaSurgery Centre, Edmonton, Alberta
  - Brunswick Dermatology Center, Fredericton, New Brunswick
  - DermEffects, London, Ontario
  - North York Research, Inc, Toronto, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
- Czechia (2):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Sanatorium Profesora Arenbergera, Prague
- Denmark (3):
  - Bispebjerg Hospital, Dermato-Venerologisk Afdeling Og Videncenter for Sårheling, D/S., Copenhagen NV
  - OUH, Odense C
  - Sjællands Universitetshospital, Roskilde
- France (4):
  - Service de dermatologie, hôpital Archet 2, CHU NICE, Nice Alpes, Maritimes
  - Hopital Edouard Herriot - CHU Lyon, Lyon
  - CHU Poitiers - Hôpital la Milétrie, Poitiers
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen
- Germany (6):
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - BAG Dr. Freitag und Knöll, Falkensee, Brandenburg
  - Klinikum Oldenburg AöR, Oldenburg, Lower Saxony
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum Carl Gustav Carus TU Dresden, Klinik und Poliklinik f. Dermatologie, Dresden, Saxony
  - Charité - Universitätsmedizin Berlin, Berlin
- Greece (6):
  - General Hospital of Athens "Evangelismos", Athens
  - 401 General Military Hospital of Athens, Athens
  - University General Hospital "Attikon", Athens
  - Andreas Syggros Hospital, Athens
  - University General Hospital of Larissa, Larissa
  - General Hospital Papageorgiou, Thessaloniki
- Poland (6):
  - Specjalistyczny Gabinet Dermatologiczny Aplikacyjno-Badawczy Marek Brzewski, Pawel Brzewski Spolka Cywilna, Krakow
  - Centrum Badawcze Panaceum Agnieszka Brzezicka Magdalena Lenkiewicz Sp. z o.o., Malbork
  - Kliniczny Szpital Wojewodzki nr 1 im.F.Chopina, Rzeszów
  - LASER CLINIC S.C. Dr Tomasz Kochanowski Dr Andrzej Krolicki, Szczecin
  - Clinical Research Group Sp. z o.o., Warsaw
  - Centralny Szpital Kliniczny MSWiA, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com